CLINICAL TRIAL: NCT01907165
Title: A Pharmacodynamic Study of Proteasome Inhibition by Disulfiram in Patients With Glioblastoma
Brief Title: Disulfiram in Treating Patients With Glioblastoma Multiforme After Radiation Therapy With Temozolomide
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201308038
Record Dates: First submitted 2013-07-19; First posted 2013-07-24 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Disulfiram; Gluconates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maintenance Temozolomide + Disulfram (Experimental): Beginning 4-6 weeks after completion of radiation therapy, patients receive maintenance temozolomide 150-200 mg/m2 PO QD on Days 1-5 every 28 days for 6 months. Disulfiram (dose level 0 = 500 mg PO QD or dose level 1 1000 mg PO QD) on days 1-28. Treatment repeats every 28 days for 6 courses* in the absence of disease progression or unacceptable toxicity.
  NOTE: *Patients may receive additional maintenance temozolomide at the discretion of the treating medical oncologist.
  Interventions: Drug: Temozolomide; Drug: Disulfiram
- Maintenance Temozolomide + Disulfiarm + Copper Gluconate (Experimental): Beginning 4-6 weeks after completion of radiation therapy, patients receive maintenance temozolomide 150-200 mg/m2 PO QD on Days 1-5 every 28 days for 6 months, disulfiram 500 mg PO QD (dose of disulfiram determined to be the MTD) on Days 1-28, and copper gluconate 6 mg PO QD on Days 1-28. Treatment repeats every 28 days for 6 courses* in the absence of disease progression or unacceptable toxicity.
  NOTE: *Patients may receive additional maintenance temozolomide at the discretion of the treating medical oncologist.
  Interventions: Drug: Temozolomide; Drug: Disulfiram; Dietary Supplement: Copper gluconate

INTERVENTIONS:
Drug: Temozolomide
  Other Names: Temodar
Drug: Disulfiram
  Other Names: Antabuse
Dietary Supplement: Copper gluconate
  Arms: Maintenance Temozolomide + Disulfiarm + Copper Gluconate

SUMMARY:
This clinical trial studies disulfiram in treating patients with glioblastoma multiforme (GBM) who have completed radiation therapy with temozolomide. Disulfiram may block some of the enzymes needed for tumor cell growth and improve clinical outcome in GBM patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically confirmed GBM (WHO grade IV).
* At least 18 years of age.
* ECOG performance status of at least 2.
* Has received or is in the process of completing a course of definitive radiotherapy of at least 45 Gy with concurrent temozolomide (patient may be registered before completing radiotherapy as long as it is anticipated that s/he will complete at least 45 Gy).
* Eligible for and planning to receive maintenance temozolomide after completion of definitive radiotherapy plus temozolomide.
* Willing to remain abstinent from consuming alcohol while on disulfiram.
* Meets the following laboratory criteria:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin > 9.0 g/dL (transfusion and/or ESA allowed)
  * Total bilirubin ≤ 2x institutional upper limit of normal (ULN)
  * AST and ALT < 3 x ULN
  * Calculated creatinine clearance must be > 60 mL/min (by Cockcroft-Gault)
* Females of childbearing potential (defined as a female who is non-menopausal or surgically sterilized) must be willing to use an acceptable method of birth control (i.e., hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to take oral medication.
* Able to understand and willing to sign an IRB-approved written informed consent document (legally authorized representative permitted).

Exclusion Criteria:

* Receipt of any other investigational agents within 14 days prior to study enrollment.
* Enrolled on another clinical trial testing a novel therapy or drug.
* History of allergic reaction to disulfiram.
* Treatment with clinically significant cytochromes P450 enzyme inducers, such as phenytoin, phenobarbital, chlordiazepoxide, diazepam, isoniazid, metronidazole, warfarin, amitriptyline within 14 days prior to the first dose of disulfiram. Of note, lorazepam and oxazepam are not affected by the P450 system and are not contraindicated with disulfiram.
* Active or severe hepatic, cardiovascular, or cerebrovascular disease, including myocardial infarction within 6 months prior to enrollment, have New York Heart Association (NYHA) Class III or IV heart failure (Appendix B), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* History of idiopathic seizure disorder, psychosis or schizophrenia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of initiation of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Pharmacological effect of disulfiram in GBM patients | 30 days
  Degree of proteasome inhibition in peripheral white blood cells and rate of complete inhibition in GBM patients using descriptive statistics

SECONDARY OUTCOMES:
Local tumor control probabilities | 2 years
  The Kaplan-Meier product-limit method will be used.
Time to tumor progression | 2 years
  Modeled using the Cox proportional hazard models.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayi Huang, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karamanakos PN. Possible role for furazolidone in the treatment of glioblastoma multiforme. J BUON. 2013 Oct-Dec;18(4):1097. No abstract available. PMID 24344045
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu